CLINICAL TRIAL: NCT01906281
Title: Adipocytokines Influence on Clinical and Ultrasonographic Inflammatory Activity in Patients With Knee Osteoarthritis
Brief Title: Influence of Adipocytokines in Osteoarthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Parc Taulí Hospital Universitari (Other)
Responsible Party: Principal Investigator, Joan Calvet Fontova, Dr, Parc Taulí Hospital Universitari
Other Study IDs: Joan01
Record Dates: First submitted 2013-07-05; First posted 2013-07-24 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Osteoarthritis, Knee; Endocrine System Diseases; Cardiovascular Risk Factors
Keywords: adipocytokines; osteoarthritis; cardiovascular risk
MeSH Terms: conditions — Osteoarthritis, Knee; Endocrine System Diseases; Osteoarthritis | interventions — Arthrocentesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — First we analyze the blood and articular fluid adipocytokines. If we can define a subset of patients characterized by a pattern of adipocytokines, genetic analysis will be performed later.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Inflammatory knee osteoarthritis: One group of patients with inflammatory condition in physical evaluation. We will make a blood analyse and arthrocentesis when synovial fluid were found in ultrasound examination. Ultrasound of affected knee and carotid artery will be performed.
  Interventions: Other: Blood analyse, arthrocentesis, ultrasound examination
- Non-inflammatory knee osteoarthritis: Patients with no inflammatory condition in physical examination. We will make a blood analyse and arthrocentesis when synovial fluid were found in ultrasound examination. Ultrasound of affected knee and carotid artery will be performed.
  Interventions: Other: Blood analyse, arthrocentesis, ultrasound examination

INTERVENTIONS:
Other: Blood analyse, arthrocentesis, ultrasound examination

SUMMARY:
Adipocytokines play an important role in joint inflammation in patients with knee osteoarthritis as measured by ultrasound and high sensitivity protein-C reactive. Adipocytokines could be the link between osteoarthritis and cardiovascular risk factors more prevalent in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 50 years old with symptomatic knee osteoarthritis.

Exclusion Criteria:

* Patients with secondary osteoarthritis of the knee
* Any other rheumatologic condition.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients over 50 years who were referred for rheumatology for symptomatic knee osteoarthritis.
Sampling Method: Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-11 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
adipocytokine level | 18 months
  We will determine the adipocytokine level at the end of inclusion period between 12-18 months

SECONDARY OUTCOMES:
Ultrasound inflammatory exploration of the knee | 18 months
  we evaluate the presence of synovial fluid with ultrasound evaluation in the visit of the patient. Ultrasound evaluation will be performed by two Rheumatologists.
Ultrasound of carotid artery | 18 months
  We will evaluate patients with ultrasound exploration in order to describe the presence of atheromatous disease in the visit of the patient
Cardiovascular risk factors | 18months
  We evaluate the prevalence of cardiovascular risk factors in the symptomatic knee osteoarthritis patients, and the relationship with adipocytokines. We will evaluate blood analyse levels of cholesterol, glycemia.

CONTACTS AND LOCATIONS:
Overall Officials: jordi Gratacos, MD Ph, Study Director — Hospital Parc Tauli
Locations (2):
- Spain (2):
  - Hospital Parc Tauli Sabadell, Sabadell, Barcelona
  - Hospital Parc Tauli, Sabadell, Barcelona